CLINICAL TRIAL: NCT06726720
Title: A Prospective, Observational, Real World Multi-cohort Study of Patients With Non-small Cell Lung Cancer (NSCLC) Initiating AstraZeneca (or Alliance Developed) Drugs
Brief Title: UmbREALung - A Retrospective and Prospective, Observational, Real World Multi-cohort Study of Patients With Non-small Cell Lung Cancer (NSCLC) Initiating Approved Drugs Developed by AZ or as Part of an AZ Alliance
Acronym: UmbREALung
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00060
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Real World Multi-cohort Study of Patients With Non-small Cell Lung Cancer (NSCLC) Initiating Approved Drugs Developed by AZ or as Part of an AZ Alliance
Keywords: observational, real world study, RWE, non-small cell lung cancer, multi-cohort, Ambispective, Prospective, Retrospective, Durvalumab, Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 - Resectable: Ambispective, observational, study of patients with non-small cell lung cancer initiating approved drugs developed by AZ or as part of an AZ alliance in resectable NSCLC
- Cohort 2 - Unresectable: Ambispective, observational, study of patients with non-small cell lung cancer initiating approved drugs developed by AZ or as part of an AZ alliance in Unresectable NSCLC
- Cohort 3 - Metastatic: Ambispective, observational, study of patients with non-small cell lung cancer initiating approved drugs developed by AZ or as part of an AZ alliance in Metastatic NSCLC

SUMMARY:
This is an ambispective, observational, multicenter and multicohort study, targeting patients with NSCLC initiating approved drugs developed by AZ or as part of an AZ alliance, in the participating countries, as monotherapy or in combination at any stage of disease. Three cohorts are designed, based on the stage of NSCLC (resectable, unresectable and metastatic). The multicohort study is modular in design. Specific modules will be set up separately to assess each new indication of drugs developed by AZ or as part of an AZ alliance once European marketing authorization (MA) has been granted and made available in the participating countries.

Patients will be enrolled in the study if they have received (retrospective), receive (retrospective and prospective) or will receive (prospective) approved drugs developed by AZ or as part of an AZ alliance according to the eligibility criteria.

Treatment plan and decision are made independently by each treating physician prior to inclusion in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* Patients with histologically or cytologically proven NSCLC
* Patients initiated with approved drugs developed by AZ or as part of an AZ alliance at the time of the enrollment or within the previous three weeks.
* Informed patients who consent to participate in the study as per local regulations.

Exclusion Criteria:

* Patients participating in an interventional clinical trial for NSCLC*

  * with the exception on low-interventional studies (RIPH2) where the intervention does not involve the NSCLC treatment
* Patients already enrolled in another module of the cohort in UMBREALUNG
* Patients under safeguard of justice, curatorship or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out with hospital and / or private clinics / hospitals (pulmonologist, medical oncologists) specialized in the treatment of patients with NSCLC in France and in Germany or any other participating countries afterwards.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Cohort A (resectable NSCLC)-Adjuvant rw DFS | 3 years
  wDFS is defined as the time from the index date (date of first administration of module specific approved drugs developed by AZ or as part of an AZ alliance) to the date of first investigator-determined recurrence (local or distant) or death (due to any cause), whichever occurs first. A patient who dies without reported recurrence will be considered to have recurred on the date of death. For patients who remain alive and whose disease has not recurred, DFS will be censored on the date of last evaluable disease assessment
Cohort A (resectable NSCLC)- Peri-operative rw EFS | 3 years
  rwEFS is defined as the time from the index date (date of first administration of module specific approved drugs developed by AZ or as part of an AZ alliance ) to the date of progression of the disease (PD) that precluded definitive surgery or discovered while attempting surgery, local or distant recurrence, or death (due to any cause), whichever occurs first. A patient who dies without reported recurrence will be considered to have event on the date of death. For patients who remain alive and who had no event, EFS will be censored on the date of last evaluable disease assessment
Cohort B (unresectable NSCLC): median rwTFST | 3 years
  real-world time to first subsequent systemic therapy (rwTFST) is defined as the time from the index date (date of first administration of module-specific approved drugs developed by AZ or as part of an AZ alliance ) to the date of first subsequent systemic therapy or the date of death (due to any cause). For patients still receiving the module-specific AZ approved drug at the end of follow-up, rwTFST will be censored on the last recorded day of ongoing treatment
Cohort C (metastatic NSCLC) rw TFST | 3 years
  real-world time to first subsequent systemic therapy (rwTFST) is defined as the time from the index date (date of first administration of module-specific approved drugs developed by AZ or as part of an AZ alliance ) to the date of first subsequent systemic therapy or the date of death (due to any cause). For patients still receiving the module-specific AZ approved drug at the end of follow-up, rwTFST will be censored on the last recorded day of ongoing treatment

SECONDARY OUTCOMES:
Response rates - all cohorts | Response evaluation via patient's best response (PR, CR, SD, PD) and date of best response
  Response is assessed via clinical or radiologic judgment or RECIST criteria
Additional rw EFS (cohort A - Peri-operative) | rw EFS and rates at 6 months, 1y, 3y, 5y (rwEFS6m, rwEFS1y, rwEFS3y, rwEFS5y)
  rwEFS is defined as the time from the index date (date of first administration of module specific approved drugs developed by AZ or as part of an AZ alliance ) to the date of progression of the disease (PD) that precluded definitive surgery or discovered while attempting surgery, local or distant recurrence, or death (due to any cause), whichever occurs first. A patient who dies without reported recurrence will be considered to have event on the date of death. For patients who remain alive and who had no event, EFS will be censored on the date of last evaluable disease assessment.
Additional rwDFS (Cohort A- adjuvant) | rwDFS and rates at 6 months, 1y, 3y, 5y (rwDFS6m, rwDFS1y, rwDFS3y, rwDFS5y)
  rwDFS is defined as the time from the index date (date of first administration of module specific approved drugs developed by AZ or as part of an AZ alliance ) to the date of first investigator-determined recurrence (local or distant) or death (due to any cause), whichever occurs first. A patient who dies without reported recurrence will be considered to have recurred on the date of death. For patients who remain alive and whose disease has not recurred, DFS will be censored on the date of last evaluable disease assessment
rwPFS (cohort B and C) | Endpoints will be median real-world Progression Free Survival (rwPFS) and rates at 6, 12, 18, 24, 36 months and 5 years (rwPFS6m, rwPFS12m, rwPF18m, rwPFS24m, rwPFS36m, rwPFS5y)
  rwPFS defined as time from index date to progression (PD) or death due to any cause.
Early progressors-rates and characteristics of patients - all cohorts | within 6 months
  Early progressors (within 6 months) based on progression-free or recurrence-free survival
rwPFS2 (all cohorts) | rwPFS2 and rates at 6, 12, 18, 24, 36 months and 5 years (rwPFS2-6m, rwPFS2-12m, rwPFS2-18m, rwD-RFS24m, rwPFS2-3y, rwPFS2-5y)
  rwPFS2 defined as time from index date to the earliest progression event subsequent to that used for the PFS endpoint or death due to any cause. Endpoints will be median time to second real-world progression (mrwPFS2) and rates
rwD-RFS or rwD-PFS ( cohort A and B) | rwD-RFS and rates at 6, 12, 18, 24, 36 months and 5 years or rwD-PFS and rates at 6, 12, 18, 24, 36 months and 5 years
  Real-word distant progression-free (rwD-PFS) or distant recurrence-free survival (rwD-RFS), defined as the time from index date to an event of distant progression or distant recurrence or death due to any cause, whichever occurred first. Endpoints will be median time to second real world to the event and rates
Real-word locoregional recurrence-free survival (rwL-RFS) - cohort A and B | rwL-RFS and rates at 6, 12, 18, 24, 36 months and 5 years (rwL-RFS6m, rwL-RFS12m, rwL-RFS18m, rwL-RFSm, rwL-RFS3y,rrwL-RFS5y)
  Real-word locoregional recurrence-free survival (rwL-RFS), defined as the time from index date to an event of local progression or local recurrence or death due to any cause, whichever occurred first. Endpoints will be median time to event and rates
rwOS - all cohorts | rwOS and rates at 6, 12, 18, 24, 36 months and 5 years (rwOS6m, rwOS12m, rwOS18m, rwOS24m, rwOS3y,rwOS5y)
  rw OS is defined as the time from the index date to death due to any cause, Real world median Endpoints will be median time to the event and rates
Real world time to treatment discontinuation (rwTTD) - all cohorts | 3 or 5 years
  rwTTD is defined as the time from the index date (date of first administration of module-specific AZ-approved drug) to the date of last administration (+duration of the drug cycle, when applicable) or date of death (due to any cause). A patient who dies without reported treatment discontinuation will be considered to have discontinued on the date of death. For patients still receiving the selected drug at the end of follow-up, TTD will be censored on the last recorded day of ongoing treatment.
Real world time to next treatment (rwTTNT) - all cohorts | rwTTNT and rates at 6 months, 1y, 3y,5y (rwTTNT6m, rwTTNT1y, rwTTNT3y,rwTTNTS5y)
  Real world time to next treatment (rwTTNT) as defined the period from the start of the treatment to the start of the next line of treatment. In the resectable cohort, local treatment will be considered as new treatment (surgery, radiotherapy) as occurring after a confirmation of progression. Endpoints will be median time to event and rates
Real world time to first subsequent local treatment (rwTFST-local treatment) all cohorts | 3 or 5 years
  Real world time to first subsequent local treatment (rwTFST-local treatment) as defined as the time from the index date (date of first administration of module specific approved drugs developed by AZ or as part of an AZ alliance ) to the date of first subsequent local therapy (including supportive or curative RT or surgery) or the date of death (due to any cause)
rwTFST (systemic) - cohort A and B | 3 or 5 years
  rwTFST is defined as the time from the index date (date of first administration of module-specific AZ-approved drug) to the date of first subsequent systemic therapy or the date of death (due to any cause). For patients still receiving the module-specific approved drugs developed by AZ or as part of an AZ alliance at the end of follow-up, rwTFST will be censored on the last recorded day of ongoing treatment
Description of associated therapies | 3 or 5 years
  Associated therapies will comprise curative therapies for NSCLC, including surgery, radiotherapy (RT), associated chemotherapy and radiotherapy (CRT), as used to treat different stages of the disease in addition to the approved drugs developed by AZ or as part of an AZ alliance subject of the specific module. Outcomes related to this objective are specific to each stage of the disease and thus to each cohort. For resectable and unresectable NSCLC (cohort A and B), the treatment of the primitive tumor will include neoadjuvant treatment, curative treatment (surgery for cohort A and CRT for cohort B) and post-curative adjuvant or consolidation treatment.
  For mNSCLC (cohort C), the treatment will describe the line of systemic treatment received (including CT) and the supportive RT or surgery when applicable.

CONTACTS AND LOCATIONS:
Locations (40):
- France (40):
  - Research Site, Aix-en-Provence
  - Research Site, Angers
  - Research Site, Aurillac
  - Research Site, Auxerre
  - Research Site, Avignon
  - Research Site, Blois
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Carcassonne
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Châteauroux
  - Research Site, Créteil
  - Research Site, Dieppe
  - Research Site, Dinan
  - Research Site, Dreux
  - Research Site, Epagny Metz Tessy
  - Research Site, Le Coudray
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Meaux
  - Research Site, Metz
  - Research Site, Mulhouse
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Neuilly-sur-Seine
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Perpignan
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Etienne
  - Research Site, Saint-Herblain
  - Research Site, Suresnes
  - Research Site, Toulouse
  - Research Site, Troyes
  - Research Site, Valenciennes
  - Research Site, Vannes
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villeurbanne

IPD SHARING:
Plan to Share IPD: No